CLINICAL TRIAL: NCT03344640
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group, Phase II, 24-week Study Investigating the Efficacy, Safety and Tolerability of AIN457 in Patients With Active Overuse Tendinopathy Refractory to Oral NSAIDs/Acetaminophen, Physiotherapy or Corticosteroid Injections
Brief Title: Study of Efficacy, Safety and Tolerability of AIN457 in Patients With Active Overuse Tendinopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457X2201; 2017-003099-30 (EudraCT Number)
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Results first posted 2020-12-09 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Tendinopathy
Keywords: Overuse tendinopathy; shoulder; rotator cuff; IL-17A-Ab; AIN457X
MeSH Terms: conditions — Tendinopathy | interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients and investigators were blinded until EOS. Sponsor was blinded until after the analysis of the primary endpoint at week 14.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- secukinumab (Experimental): AIN457 300 mg subcutaneously (s.c.) for 12 weeks
  Interventions: Drug: secukinumab
- Placebo (Placebo Comparator): Placebo subcutaneously for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: secukinumab — AIN457 300 mg subcutaneously for 12 weeks
  Other Names: AIN457
  Arms: secukinumab
Other: Placebo — Placebo to match AIN457 subcutaneously for 12 weeks
  Arms: Placebo

SUMMARY:
This was a randomized, double-blind, placebo-controlled, multi-center, Phase II study of s.c. secukinumab 300 mg in 98 randomized patients with overuse rotator-cuff tendinopathy without systemic inflammatory disease.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled, multi-center, Phase II study of s.c. secukinumab 300 mg in 98 randomized patients with overuse rotator-cuff tendinopathy without systemic inflammatory disease and refractory to NSAIDs/acetaminophen, physiotherapy or corticosteroids.

The study consisted of a 4-week screening period, a 2-week run-in period, a 12-week treatment period and a 12-week follow-up period after last treatment. The population consisted of patients with unilateral overuse (non-systemic inflammatory) shoulder tendinopathy, 18 - 65 years of age.

Safety assessments included physical examinations, ECGs, vital signs, standard clinical laboratory evaluations (hematology, blood chemistry, and urinalysis), adverse event and serious adverse event monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female patients 18 to 65 years of age at randomization
2. Presence of unilateral rotator cuff tendinopathy with:

   1. Symptoms present ≥6 weeks, but <12 months prior to randomization
   2. Tendinopathy with no more than a 50% tear as established by ultrasound at screening (historic data acceptable if not older than 3 months) and MRI at baseline: Sein MRI tendinopathy scoring system grade I-III; with no tear or partial tear [maximum 50% tendon thickness (Bauer tendon thickness score maximum 2); AP length maximum 10 mm (Bauer tendon length score max 2)]. Maximum 50% of patients with partial tear
   3. Pain in the affected shoulder (at rest or on movement) on at least 3 days out of 7 days in the past week prior to baseline and a score of ≥4 out of 10 on a VAS pain scale
   4. Positive "Painful Arc Test" on examination and/or nightly pain in the affected shoulder on at least 4 out of 7 days in the past week prior to baseline
3. The rotator-cuff tendinopathy must have been refractory to standard treatment, including NSAIDs and physiotherapy

Exclusion Criteria:

1. Rheumatologic, inflammatory diseases, including but not limited to: PsA, AS and RA 2. Previous shoulder surgery in affected shoulder 3. History of adhesive capsulitis/frozen shoulder or calcification in the tendon (in affected or contralateral shoulder) confirmed by X-Ray, historic X-Rays can be used if performed within 3 months of baseline 4. Symptomatic osteoarthritis of the shoulder (gleno-humeral, acromioclavicular) (in affected or contralateral shoulder confirmed by X-Ray, historic X-Rays can be used if performed within 3 months of baseline 5. Neck conditions, including but not limited to cervical spine syndrome, which in the opinion of the investigator, may explain the patient's symptoms 6. Previous platelet rich plasma injections within the last 12 months prior to randomization 7. Previous treatment with any cell-depleting therapies including but not limited to anti- CD20, investigational agents (e.g. Campath, anti-CD4, anti-CD5, anti-CD3, anti-CD19) 8. Previous exposure to any biologic immunomodulating agents, including but not limited to TNFalpha inhibitors (including, but not limited to adalimumab, infliximab), or biologics targeting IL-17 (including, but not limited to secukinumab, ixekizumab or brodalumab) or the IL-17 receptor within the last 12 months prior to baseline 9. Any intraarticular/subacromial corticosteroid treatment within 8 weeks prior to randomization and more than 3 injections for the current tendinopathy. Oral, intramuscular or i.v. corticosteroid treatment within the last 12 months prior to randomization

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (5):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, La Mesa, California
  - Novartis Investigative Site, Clearwater, Florida
  - Novartis Investigative Site, Miami Lakes, Florida
  - Novartis Investigative Site, Tampa, Florida
- Czechia (3):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Kolín, Czech Republic
  - Novartis Investigative Site, Prague
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg
- Novartis Investigative Site, Leiden, Netherlands
- Novartis Investigative Site, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=687

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of all patients randomized (N= 98; 100%) in the study, a total of 96 patients (98%) were dosed (49 patients in the secukinumab 300 mg group and 47 patients in the placebo group)
Pre-assignment Details: 2 patients were not dosed, one patient decided to discontinue on Day 1 due to a common cold and one patient was a run-in failure
Groups:
- Secukinumab: AIN457 300 mg subcutaneously (s.c.)
- Placebo: Placebo s.c.
Period: Overall Study
Arm/Group | Secukinumab | Placebo
Started | 49 | 47
Completed | 46 | 44
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2
Period: Follow-up Epoch
Arm/Group | Secukinumab | Placebo
Started | 46 | 44
Completed | 46 | 42
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAS) included all subjects that received any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab | Placebo | Total
Number analyzed (Participants) | 49 | 47 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] — Demographic summary (Safety analysis set)
  years | 44.8 (11.51) | 49.1 (10.56) | 46.9 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants] — 41.7% of participants were female, and 58.3% were male
  Participants
    Female | 17 | 23 | 40
    Male | 32 | 24 | 56
Race/Ethnicity, Customized [Number; unit: Participants] — 1% Asian, 4.2% Black or African American, 91.7% White, 1% Unknown, 2.1% Other
  Participants
    Asian | 1 | 0 | 1
    Black or African American | 3 | 1 | 4
    White | 43 | 45 | 88
    Unknown | 1 | 0 | 1
    Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: The Western Ontario Rotator Cuff (WORC) Patient Reported Outcome (PRO) Score at Week 14 in All Patients - Statistical Analysis Results of Total WORC Scores at Week 14
Description: WORC PRO score at week 14. The WORC Index consists of 21 items divided into 5 Domains: Physical Symptoms (6 items), Sport/Recreation (4 items), Work Function (4 items), Lifestyle Function (4 items) and Emotional Function (3 items). The total scores and sub scores used were the percentages of the normal scores with 0 being worst and 100 being best.
  All Patients - Statistical analysis results of WORC scores at Week 14
Time Frame: Week 14 (Day 99)
Population: Pharmacodynamic (PD) Analysis Set
Measure: Number (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 47 | 41
Scores on a scale | 37.00 [30.10 to 43.90] | 37.77 [30.40 to 45.15]
Statistical Analysis 1: Comparison: Secukinumab vs Placebo; All Patients at day 99; Test type: Superiority; p = 0.875, LS mean; LS mean change from baseline in WORC total percentage score; Mean Difference (Final Values) = -0.77, 90% CI 2-sided [-8.84 to 7.30]

2. Secondary Outcome: The Western Ontario Rotator Cuff (WORC) Patient Reported Outcome (PRO) Scores Over Time in All Patients
Description: WORC score at Days 15, 29, 57, 85, 127, and End of Study (day 169). The scale range for WORC total score is 0-100, 0 being the worst possible outcome (highly symptomatic patient) and 100 being the best possible outcome (asymptomatic patient)
Time Frame: Days 15, 29, 57, 85, 127, and End of Study
Population: PD Analysis Set
Measure: Number (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 47 | 41
Scores on a scale
  Day 15 | 12.39 [6.99 to 17.79] | 8.42 [2.66 to 14.18]
  Day 29 | 22.35 [16.38 to 28.32] | 19.49 [13.11 to 25.86]
  Day 57 | 28.74 [22.19 to 35.29] | 30.11 [23.08 to 37.13]
  Day 85 | 34.86 [28.18 to 41.53] | 33.48 [26.35 to 40.61]
  Day 127 | 41.86 [34.96 to 48.77] | 38.50 [31.12 to 45.88]
  End of Study | 43.41 [36.21 to 50.61] | 40.97 [33.27 to 48.66]
Statistical Analysis 1: Comparison: Secukinumab vs Placebo; All patientts at day 15; Test type: Superiority; p = 0.190, LS mean; LS mean change from baseline in WORC total percentage score; Difference and 90% CI versus placebo = 3.97, 90% CI 2-sided [-1.03 to 8.97]
Statistical Analysis 2: Comparison: Secukinumab vs Placebo; All patients at day 29; Test type: Superiority; LS Mean; LS mean change from baseline in WORC total percentage score; Difference and 90% CI versus placebo = 3.97, 90% CI 2-sided [-3.39 to 9.11]
Statistical Analysis 3: Comparison: Secukinumab vs Placebo; All patients at day 57; Test type: Superiority; p = 0.761, LS Mean; LS mean change from baseline in WORC total percentage score; Difference and 90% CI versus placebo = 0.761, 90% CI 2-sided [-8.81 to 6.08]
Statistical Analysis 4: Comparison: Secukinumab vs Placebo; All patients at day 85; Test type: Superiority; p = 0.765, LS Mean; LS mean change from baseline in WORC total percentage score; Difference and 90% CI versus placebo = 0.765, 90% CI 2-sided [-6.27 to 9.03]
Statistical Analysis 5: Comparison: Secukinumab vs Placebo; All patients at day 127; Test type: Superiority; p = 0.491, LS Mean; LS mean change from baseline in WORC total percentage score; Difference and 90% CI versus placebo = 0.491, 90% CI 2-sided [-4.73 to 11.45]
Statistical Analysis 6: Comparison: Secukinumab vs Placebo; All patients at end of study; Test type: Superiority; p = 0.639, LS Mean; LS mean change from baseline in WORC total percentage score; Difference and 90% CI versus placebo = 2.44, 90% CI 2-sided [-6.19 to 11.07]

3. Secondary Outcome: Disability of Arm, Shoulder and Hand Questionnaire Score (QuickDASH) Over Time
Description: Patient Reported Outcome: Disability of Arm, Shoulder and Hand (QuickDASH) This questionnaire asks about symptoms as well participant's ability to do certain activities - ranging from 1 (No difficulty) to 5 (Unable).
  The scale range for QuickDASH total score is 0-100, 0 being the best possible outcome and 100 being the worst possible outcome
Time Frame: Days 15, 29, 57, 85, 99, 127, and End of Study
Population: PD Analysis Set
Measure: Number (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 47 | 41
Scores on a scale
  Day 15 | -11.64 [-16.14 to -7.14] | -8.23 [-13.02 to -3.44]
  Day 29 | -18.31 [-23.20 to -13.41] | -16.95 [-22.18 to -11.73]
  Day 57 | -22.43 [-27.55 to -17.30] | -24.01 [-29.49 to -18.52]
  Day 85 | -28.14 [-33.55 to -22.73] | -27.22 [-32.98 to -21.45]
  Day 99 | -29.45 [-34.72 to -24.19] | -30.69 [-36.30 to -25.07]
  Day 127 | -32.86 [-38.26 to -27.46] | -31.99 [-37.75 to -26.23]
  End of Study | -33.89 [-39.27 to -28.50] | -35.40 [-41.13 to -29.67]
Statistical Analysis 1: Comparison: Secukinumab vs Placebo; Statistical analysis results of QuickDASH total score (PD Analysis Set) at day 99; Test type: Superiority; p = 0.735, LS Mean — Difference and 90% CI versus placebo; LS mean change from baseline in QuickDASH total score; Difference and 90% CI versus Placebo = 1.23, 90% CI 2-sided [-4.81 to 7.28]
Statistical Analysis 2: Comparison: Secukinumab vs Placebo; Statistical analysis results of QuickDASH total score (PD analysis set) at End of Study; Test type: Superiority; p = 0.689, LS Mean; LS mean change from baseline in QuickDASH total score; Difference and 90% CI versus Placebo = 1.51, 90% CI 2-sided [-4.76 to 7.79]

4. Secondary Outcome: American Shoulder and Elbow Surgeons (ASES) Score Over Time
Description: Patient Reported Outcome: American Shoulder and Elbow Surgeons Shoulder Evaluation Form (ASES) score is self-administered and has 17 questions in the areas of shoulder symptoms and functions. The ASES total score ranges from 0 to 100 (best).
Time Frame: Days 15, 29, 57, 85, 99, 127, and End of Study
Population: PD Analysis Set
Measure: Number (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 47 | 41
Scores on a scale
  Day 15 | 8.66 [3.98 to 13.33] | 5.26 [0.26 to 10.25]
  Day 29 | 17.53 [12.35 to 22.71] | 14.37 [8.82 to 19.92]
  Day 57 | 24.15 [18.34 to 29.96] | 22.56 [16.31 to 28.81]
  Day 85 | 30.50 [24.51 to 36.50] | 26.97 [20.51 to 33.43]
  Day 99 | 31.29 [25.28 to 37.31] | 27.79 [21.33 to 34.26]
  Day 127 | 34.92 [28.80 to 41.05] | 32.94 [26.33 to 39.56]
  End of Study | 37.29 [30.97 to 43.62] | 36.15 [29.33 to 42.97]
Statistical Analysis 1: Comparison: Secukinumab vs Placebo; Statistical analysis results of ASES total score (PD analysis) at day 99; Test type: Superiority; p = 0.411, LS Mean; LS mean change from baseline in ASES total percentage score; Difference and 90% CI vesus placebo = 3.50, 90% CI 2-sided [-3.54 to 10.54]
Statistical Analysis 2: Comparison: Secukinumab vs Placebo; Statistical analysis results of ASES total score (PD analysis) at End of Study set); Test type: Superiority; p = 0.804, LS Mean; LS mean change from baseline in ASES total percentage score; Difference and 90% CI versus placebo = 1.14, 90% CI 2-sided [-6.50 to 8.78]

5. Secondary Outcome: Your Health Today Score Over Time
Description: Patient Reported Outcome: Statistical analysis results of EQ-5D-5L for Your health Today questionnaire, which reflects how good or bad the subjets Health is on a scale from 0 (worst health) to 100 (best health).
Time Frame: Days 15, 29, 57, 85, 99, 127, and End of Study
Population: PD Analysis Set
Measure: Number (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 47 | 41
Scores on a scale
  Day 15 | -0.22 [-4.02 to 3.58] | 0.02 [-4.02 to 4.07]
  Day 29 | 3.27 [-0.71 to 7.25] | 3.56 [-0.69 to 7.81]
  Day 57 | 3.19 [-1.07 to 7.45] | 9.02 [4.45 to 13.59]
  Day 85 | 7.36 [2.84 to 11.89] | 7.79 [2.96 to 12.62]
  Day 99 | 8.75 [4.13 to 13.38] | 10.01 [5.09 to 14.94]
  Day 127 | 9.55 [5.29 to 13.80] | 13.59 [9.05 to 18.13]
  End of Study | 10.22 [4.84 to 15.60] | 12.13 [6.36 to 17.89]
Statistical Analysis 1: Comparison: Secukinumab vs Placebo; Statistical analysis results of Your Health Today EQ-5D-5L Index score at day 99 (PD Analysis Set); Test type: Superiority; p = 0.706, LS Mean; LS Mean change from baseline in Your Health Today Score at day 99; Difference and 90% CI versus placebo = -1.26, 90% CI 2-sided [-6.81 to 4.29]
Statistical Analysis 2: Comparison: Secukinumab vs Placebo; Statistical analysis results of Your Health Today EQ-5D-5L Index score at End of Study; Test type: Superiority; p = 0.647, LS Mean; LS mean change from baseline in Your Health Today score; Difference and 90% CI versus placebo = -1.90, 90% CI 2-sided [-8.79 to 4.99]

6. Secondary Outcome: EQ-5D-5L Index Score Over Time
Description: Patient Reported Outcome: Statistical analysis results of EQ-5D-5L Index score, which contains 5 items to assess Health Status (mobility, self-care, usual activity, pain/discomfort, and anxiety/depression). Overall scores range from 0 to 1 with lower scores representing a higher level of dysfunction.
Time Frame: Days 15, 29, 57, 85, 99, 127 and End of Study
Population: PD Analysis Set
Measure: Number (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 47 | 41
Scores on a scale
  Day 15 | 0.07 [0.05 to 0.10] | 0.04 [0.01 to 0.07]
  Day 29 | 0.10 [0.07 to 0.13] | 0.09 [0.05 to 0.12]
  Day 57 | 0.12 [0.09 to 0.15] | 0.11 [0.08 to 0.15]
  Day 85 | 0.16 [0.13 to 0.19] | 0.14 [0.10 to 0.18]
  Day 99 | 0.16 [0.13 to 0.20] | 0.15 [0.11 to 0.19]
  Day 127 | 0.19 [0.15 to 0.23] | 0.17 [0.13 to 0.21]
  End of Study | 0.19 [0.16 to 0.23] | 0.18 [0.14 to 0.22]
Statistical Analysis 1: Comparison: Secukinumab vs Placebo; Statistical analysis results of of EQ-5D-5L Index score at day 99 (PD Analysis Set); Test type: Superiority; p = 0.613, LS Mean; LS mean change from baseline in EQ-5D-5L Index score; Difference and 90% CI versus placebo = 0.01, 90% CI 2-sided [-0.03 to 0.06]
Statistical Analysis 2: Comparison: Secukinumab vs Placebo; Statistical analysis results of of EQ-5D-5L Index score at End of Study (PD Analysis Set); Test type: Superiority; p = 0.740, LS Mean; LS mean change from baseline in EQ-5D-5L Index score; Difference and 90% CI versus placebo = 0.02, 90% CI 2-sided [-0.04 to 0.06]

7. Secondary Outcome: Pain Score Over Time Using a VAS Scale
Description: Pain intensity is assessed by a Visual Analog Scale (VAS) which is measured on a 100mm line that represents a continuum between "no pain" and "worst pain".
  The scale range for pain score is 0-100, 0 being the best possible outcome (no pain) and 100 being the worst possible outcome (worst pain).
Time Frame: Days 15, 29, 57, 85, 99, 127 and End of Study
Population: PD Analysis Set
Measure: Number (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 47 | 41
Scores on a scale
  Day 15 | -12.11 [-19.52 to -4.70] | -9.50 [-17.30 to -1.71]
  Day 29 | -26.04 [-33.97 to -18.11] | -23.13 [-31.52 to -14.74]
  Day 57 | -35.52 [-43.67 to -27.37] | -32.83 [-41.52 to -24.15]
  Day 85 | -42.63 [-50.88 to -34.38] | -37.97 [-46.74 to -29.21]
  Day 99 | -46.11 [-54.10 to -38.12] | -40.56 [-49.00 to -32.11]
  Day 127 | -49.44 [-57.45 to -41.44] | -45.27 [-53.75 to -36.79]
  End of Study | -52.23 [-60.31 to -44.14] | -50.74 [-59.40 to -42.08]
Statistical Analysis 1: Comparison: Secukinumab vs Placebo; Statistical analysis results of pain score using VAS scale (PD Analysis Set) at day 99; Test type: Superiority; p = 0.281, LS Mean; LS MMean CFB (90% CI); Difference and 90% CI versus placebo = -5.55, 90% CI 2-sided [-14.07 to 2.97]
Statistical Analysis 2: Comparison: Secukinumab vs Placebo; Statistical analysis results of pain score using VAS scale (PD Analysis Set) at End of Study; Test type: Superiority; p = 0.780, LS Mean; LS Mean CFB (90% CI); Difference and 90% CI versus placebo = -1.49, 90% CI 2-sided [-10.33 to 7.35]

8. Secondary Outcome: Patient Global Assessment (PGA) Score Over Time Using a VAS Scale
Description: The patient's global assessment of disease activity is performed using a 100 mm Visual Analog Scale (VAS) ranging from "no activity" to "most active" in the last 24 hours.
  The scale range for PGA score is 0-100, 0 being the best possible outcome (no disease activity) and 100 being the worst possible outcome (maximal disease activity).
Time Frame: Days 15, 29, 57, 85, 99, 127 and End of Study
Population: PD Analysis Set
Measure: Number (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 47 | 41
Scores on a scale
  Day 15 | -6.33 [-13.44 to 0.79] | -8.09 [-15.79 to -0.38]
  Day 29 | -22.25 [-29.68 to -14.82] | -16.38 [-24.43 to -8.33]
  Day 57 | -29.40 [-37.06 to -21.74] | -25.69 [-34.04 to -17.34]
  Day 85 | -37.57 [-45.01 to -30.12] | -31.75 [-39.79 to -23.72]
  Day 99 | -38.43 [-45.88 to -30.97] | -35.10 [-43.14 to -27.07]
  Day 127 | -43.78 [-51.23 to -36.33] | -38.32 [-46.37 to -30.26]
  End of Study | -47.72 [-55.15 to -40.28] | -39.43 [-47.45 to -31.40]
Statistical Analysis 1: Comparison: Secukinumab vs Placebo; Statistical analysis results of pain score using VAS scale (PD Analysis Set) at day 99; Test type: Superiority; p = 0.489, LS Mean; LS Mean change from baseline in VAS score; Difference and 90% CI versus placebo = -3.32, 90% CI 2-sided [-11.28 to 4.64]
Statistical Analysis 2: Comparison: Secukinumab vs Placebo; Statistical analysis results of pain score using VAS scale at End of Study; Test type: Superiority; p = 0.087, LS Mean; LS Mean change from baseline in VAS score; Difference and 90% CI versus placebo = -8.29, 90% CI 2-sided [-16.26 to -0.32]

9. Secondary Outcome: Physician Global Assessment (PhGA) Score Using a VAS Scale Over Time
Description: Physician global assessment (PhGA) score using a VAS scale (considering the last 24 hours).
  The scale range for PhGA score is 0-100, 0 being the best possible outcome (no disease activity) and 100 being the worst possible outcome (maximal disease activity).
Time Frame: Days 15, 29, 57, 85, 99, 127 and End of Study
Population: PD Analysis Set
Measure: Number (90% Confidence Interval); unit: Score on a scale
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 47 | 41
Score on a scale
  Day 15 | -13.99 [-20.22 to -7.75] | -9.11 [-15.80 to -2.42]
  Day 29 | -25.01 [-31.51 to -18.50] | -19.42 [-26.42 to -12.43]
  Day 57 | -30.78 [-37.57 to -23.99] | -27.83 [-35.13 to -20.53]
  Day 85 | -33.42 [-40.68 to -26.16] | -37.88 [-45.66 to -30.11]
  Day 99 | -35.72 [-42.66 to -28.79] | -41.73 [-49.15 to -34.31]
  Day 127 | -41.72 [-48.32 to -35.12] | -44.18 [-51.28 to -37.08]
  End of Study | -44.64 [-51.86 to -37.41] | -44.26 [-52.02 to -36.51]
Statistical Analysis 1: Comparison: Secukinumab vs Placebo; Statistical analysis results of PhGA score using VAS scale at day 99; Test type: Superiority; p = 0.210, LS Mean; LS Mean CFB (90% CI); Difference and 99% CL versus placebo = 6.10, 90% CI 2-sided [-1.90 to 13.91]
Statistical Analysis 2: Comparison: Secukinumab vs Placebo; Statistical analysis results of PhGA score using VAS scale at End of Study; Test type: Superiority; p = 0.942, LS Mean; LS Mean CFB (90% CI); Difference and 90% CI versus placebo = -0.37, 90% CI 2-sided [-8.86 to 8.11]

10. Secondary Outcome: Pharmacokinetics - Cmin
Description: Mean trough concentrations
  Cmin is a pharmacokinetics term for the minimum blood plasma concentration reached by a drug prior to administration of a second dose (mass/volume)
  Serum trough concentrations of secukinumab 300 mg group was measured at Days 1, 29, 85 and EoS
Time Frame: Days 1, 29, 85 and EoS (End of Study)
Population: PD Analysis Set
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Secukinumab
Number analyzed (Participants) | 47
ug/mL
  Mean trough concentration after first 4 wkly doses | 90.4 (30.7)
  Week 12 | 13.2 (6.67)

11. Secondary Outcome: Immunogenicity Assessment - Treatment Emergent ADAs
Description: Number of Participants with Treatment emergent Anti-secukinumab antibodies
Time Frame: Day 1 and EoS
Population: PD Analysis Set
Measure: Number; unit: Participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 47 | 41
Participants
  Day 1 | 0 | 1
  End of Study | 0 | 0

12. Secondary Outcome: Number of Participants With Tendinosis Grade Score 1, 2 or 3 Measured by Magnetic Resonance Imaging (MRI) Sein Scores
Description: Assessment of structural changes in the rotator cuff tendinopathy over time
  The MRI Sein score was used to grade supraspinatus tendinosis using a modified 4-point scale from 0 to 3 and changes in grading over time were captured in the shift table. Grade 0 is normal, grade 1 is mild, Grade 2 is moderate and grade 3 is marked tendinosis.
  In this Sein score assessment, only data from Day 99 and baseline could be compared, as only those two time points were double read and adjudicated in case the 2 readers had different results. At any other time-points (Day 57 and EOS), images were assessed only by one reader and thus could not be compared to baseline.
Time Frame: Baseline and Day 99
Population: PD Analysis Set
Measure: Number; unit: participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 47 | 41
participants
  Baseline grade 1 | 31 | 25
  Baseline grade 2 | 11 | 10
  Baseline grade 3 | 3 | 3
  Day 99 grade 1 | 31 | 26
  Day 99 grade 2 | 11 | 9
  Day 99 grade 3 | 3 | 3

ADVERSE EVENTS:
Time Frame: Approximately 40 weeks: 15 Dec 2017 through 17 Oct 2019
Description: Adverse Events (AEs) are any untoward sign or symptom that occurs during the study treatment
Groups:
- AIN457 300 mg s.c.: AIN457 300 mg
Arm/Group | AIN457 300 mg s.c. | Placebo
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/47
Other Adverse Events (participants affected / at risk) | 36/49 | 34/47
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 300 mg s.c. (N=49) | Placebo (N=47)
Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Faeces soft (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 5
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 2
Feeling hot (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Injection site erythema (General disorders) | 1 | 2
Injection site haematoma (General disorders) | 2 | 1
Injection site pain (General disorders) | 0 | 1
Injection site paraesthesia (General disorders) | 1 | 0
Injection site pruritus (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 0 | 1
Acute sinusitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1
Fungal skin infection (Infections and infestations) | 3 | 0
Gastroenteritis (Infections and infestations) | 2 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1
Gastrointestinal viral infection (Infections and infestations) | 1 | 0
Lymphangitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 8 | 5
Oral candidiasis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0
Periodontitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pulpitis dental (Infections and infestations) | 0 | 1
Pustule (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 4
Urinary tract infection (Infections and infestations) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Injection related reaction (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Red blood cell sedimentation rate increased (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Benign bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1
Dizziness postural (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 7 | 7
Paraesthesia (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Phonophobia (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Keratolysis exfoliativa acquired (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
In general "End of Study" is Day 169 (week 24). But in the study it was handled in a way, that whenever a subject discontinued the last visit was the EoS visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety

DOCUMENTS (2):
  • Study Protocol (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/40/NCT03344640/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT03344640/SAP_001.pdf